CLINICAL TRIAL: NCT04189029
Title: Redefining the Phenotypic Spectrum of Heart Failure With Preserved Ejection Fraction (HFpEF) by Deep Phenotyping and Machine Learning Methods: The PACIFIC-PRESERVED Study (PhenomApping, ClassIFication, and Innovation for Cardiac Dysfunction - HF With PRESERVED LVEF Study)
Brief Title: PACIFIC-PRESERVED : PhenomApping, ClassIFication, and Innovation for Cardiac Dysfunction - HF With PRESERVED LVEF Study
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: BPIfrance (Other); Sanofi (Industry); Institut de Recherches Internationales Servier (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); BioSerenity (Industry); Casis (Unknown); Firalis SA (Industry); Fealinx (Unknown); Centre National de la Recherche Scientifique, France (Other); ESPCI Paris (Other); University of Paris 5 - Rene Descartes (Other); Sorbonne University (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190558; 2019-A01795-52 (Other: N° IDRCB)
Record Dates: First submitted 2019-11-28; First posted 2019-12-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma, Serum, PaxGene RNA, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF patients: Heart failure patients (NYHA II-IV) with left ventricular ejection fraction ≥ 50%, 1000 patients anticipated among which up to 300 with extensive phenotyping
  Interventions: Other: Extensive phenotyping
- HFrEF patients: Heart failure patients (NYHA II-IV) with left ventricular ejection fraction ≤ 40%, 1000 patients anticipated among which up to 100 with extensive phenotyping (age- and gender-matched on participating HFpEF patients)
  Interventions: Other: Extensive phenotyping
- Subjects apparently without heart failure: Subjects without history or signs of heart failure, up to 100 subjects anticipated with extensive phenotyping (age- and gender-matched on participating HFpEF patients)
  Interventions: Other: Extensive phenotyping

INTERVENTIONS:
Other: Extensive phenotyping — Prospective assessment of physical evaluation, biomarkers and omics, cardiac and vascular imaging and telemonitoring of cardiovascular parameters for 14 days.

SUMMARY:
This is a prospective multicenter study to decipher phenotypic variability within patients with heart failure and preserved left ventricular ejection fraction (HFpEF). From a registry of heart failure patients (2500 anticipated) hospitalized in the participating centers in the last 3 years, up to 300 participants (with a final ratio of 3 HFpEF patients, 2 patients with heart failure and reduced ejection fraction (HFrEF) and 1 matched subjects without heart failure will be enrolled for an extensive phenotyping with physical evaluation, biomarkers and omics, cardiac and vascular imaging and telemonitoring of cardiovascular parameters. Cluster analysis with machine learning methods will be performed to define phenogroups unique to the HFpEF patient population.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a complex and prevalent syndrome with currently no efficient therapy. This syndrome is likely explained by different pathophysiological inputs leading to common symptoms of heart failure. These pathophysiological abnormalities can primarily involve the heart but also other organs with secondary impact on the myocardium. There is however no clear understanding and diagnostic algorithms of the different HFpEF subpopulations. Novel mathematical methods (such as machine learning) can help identifying clusters within an heterogeneous population such as HFpEF patients.

A registry (2500 anticipated) will be constituted with patients hospitalized for congestive heart failure in the participating centers during the last 3 years. From this registry, up to 500 patients will be invited to visit in the hospital for 8-10 hours for physical examination, ECG, performance-based tests, blood draw, cMRI, echocardiography (rest and low-level exercise), Ultrafast echo (for non-invasive measurement of myocardial stiffness), low radiation cardiac CT (for calcium scoring), non-invasive measurement of arterial stiffness. They will be asked to fill out questionnaires about dyspnea, depression and about general health and quality of life. They will then be equipped with a smart connected garment (with cardiovascular & hemodynamic sensors), a connected weight balance and a blood pressure monitoring device for telemonitoring collection of cardiovascular hemodynamic parameters in real-life conditions (for 14 days).

Patients included in the registry will be followed-up for 3 years using medico-administrative databases and vital status, cardiovascular and heart failure outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Affiliation to a social security scheme, universal medical coverage (CMU) or any equivalent scheme
* Physical state compatible with the carrying out of the investigations according to the judgment of the investigator
* Procedure for obtaining consent

For HFpEF patients:

* Hospitalization in one of the partner hospitals in the last 30 months
* With a diagnosis of symptomatic congestive heart failure (NYHA II to IV)
* With a plasma concentration of BNP ≥ 100 μg / ml or NT-proBNP ≥ 300 μg / ml or having had an administration of a dose of intravenous diuretics during hospitalization for congestive heart failure
* Left ventricular ejection fraction ≥ 50%
* Hospital discharge for at least 2 months

For HFrEF patients:

* Hospitalization in one of the partner hospitals in the last 30 months
* With a diagnosis of symptomatic congestive heart failure (NYHA II to IV)
* Plasma concentration of BNP ≥ 100 μg / ml or NT-proBNP ≥ 300 μg / ml or administered a dose of intravenous diuretics during hospitalization for congestive heart failure
* Hospital discharge for at least 2 months
* Left ventricular ejection fraction ≤ 40%
* Matched age and sex to HFpEF patients (for participants to extensive phenotyping)

For subjects apparently without heart failure :

* Subject without a notable medical history or medical history within the last 5 years
* Normotensive or who may have an essential hypertension of grade 1 (≤159 / 99 mmHg), treated or not
* Can present a dyslipidemia, treated by hygieno-dietetic measures alone
* Sinus heart rate
* Estimated glomerular filtration rate ≥ 60 ml / min (CKD epi)
* Matched age and sex to HFpEF patients (for participants to extensive phenotyping)

Exclusion Criteria:

All subjects

* Pregnancy or breastfeeding
* Participation in another interventional study
* Person placed under the safeguard of justice
* Subject that can not understand the procedures related to the protocol
* Severe obesity (BMI > 40 Kg / m2)
* For those performing the injected MRI: Patient who has already had a severe allergy to gadolinium MRI contrast agents
* For those performing the injected MRI: MRI usual contraindications: Pace-maker, defibrillator, metallic objects
* Administration of a vaccine dose (including anti-Sars-Cov-2) less than 3 weeks old

For both HFpEF and HFrEF patients:

* History of right ventricular infarction
* History of cardiac transplantation or circulatory assistance
* Major surgery scheduled for less than 6 months, coronary revascularization of less than 3 months
* Pacemaker or any implanted device (or foreign body) not compatible with MRI
* Presence of very severe co-morbidity: end-stage renal failure (GFR <15ml / min), severe chronic obstructive pulmonary disease (COPD), severe valve disease (including severe aortic stenosis), organ transplantation
* Hypertrophic cardiomyopathy of known genetic cause
* Hereditary amyloidosis with disabling neuropathy
* Amyloidosis under specific treatment
* Other antecedent of known congenital heart disease type, Post-embolic chronic pulmonary heart, Restrictive Cardiopathy, Diagnosed Fabry Disease

For HFpEF patients:

- History of systolic dysfunction with proven LVEF reduction (≤ 40%)

For subjects apparently without heart failure :

* Medication use other than pure systemic or local estrogen / progestin and progestin contraceptives and paracetamol, at the discretion of the investigator
* Acute pathology within 8 days prior to inclusion
* Cardiac or vascular organic impairment or apparent chronic diseases
* Chronic treatment outside a treatment for high blood pressure
* Having already had ≥3 MRI with injection of gadolinium contrast agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with different forms of heart failure (ie with preserved left ventricular ejection fraction vs. reduced left ventricular ejection fraction) and subjects apparently without heart failure
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Machine learning algorithm to identify distinct phenotypic subgroups among HFpEF patients | 14 days
  Machine learning-based cluster analysis using extensive phenotyping data from HFpEF, HFrEF and subjects without apparent HF

SECONDARY OUTCOMES:
Prognosis | 3 years
  Identify phenotypic subgroup(s) with higher risk of cardiovascular and HF outcomes
Myocardial stiffness | 3 years
  Assess the diagnostic and prognostic value of myocardial stiffness measured with ultrafast cardiac echography
Sarcopenia and muscular capacity | 3 years
  Prevalence and importance of muscle loss, weakness measured with hand grip strength test (Kg) and with the short physical performance battery (SPPB, combining the results of gait speed, chair stand and balance tests) in HFpEF patients
Exercise tolerance | 3 years
  Measure exercise tolerance with 6-minute walk test
Cardiac fibrosis | 3 years
  Prevalence, diagnostic and prognostic importance of cardiac fibrosis (as estimated by cMRI and specific biological markers) in HFpEF patients
Arterial Stiffness | 3 years
  Assess the diagnostic and prognostic value of arterial stiffness measured by pulse wave velocity
Right heart and pulmonary circulation | 3 years
  Assess the diagnostic and prognostic value of novel markers to quantify right heart function and pulmonary circulation measured with cMRI
Ventricular-arterial coupling | 3 years
  Machine learning-based analysis on 4D MRI recordings to estimate ventricular-arterial coupling
Omics signature | 3 years
  Apply multi-omics techniques (including measurements of miRNA, lNcRNA, inflammation markers, and DNA methylation level) to define specific biological signatures to HF and HFpEF patients
Quality of life evaluation | 3 years
  General and HF QOL questionnaires: Kansas city cardiomyopathy questionnaire - the sum of responses from all 12 items, Range for subscale is 0-100 and the range for the summary score is 0-100 with lower scores indicating more significant disease impact; Global quality of life score with SF36 (Short form 36 health survey): The norm data is 0-100, the health related quality of life is increased as the scores are increased.
Telemonitoring of weight | 3 years
  Remote measurement of body weight
Telemonitoring of cardiac rythm | 3 years
  Remote measurement of cardiac arrhythmias
Telemonitoring of ECG | 3 years
  Remote measurement of heart rate variability
Telemonitoring of physical activity | 3 years
  Remote measurement of physical activity with an actimeter
Telemonitoring of blood pressure | 3 years
  Remote measurements of blood pressure in mmHg
Telemonitoring of pulmonary function | 3 years
  Remote measurement of respiratory rate
Telemonitoring of oxygen saturation | 3 years
  Remote measurement of oxygen saturation (%)
Telemonitoring of pulmonary congestion | 3 years
  Remote evaluation of pulmonary congestion with measurement of thoracic impedance
Digitalized ECG | 3 years
  Develop novel machine learning based markers of HF, of HFpEF and HFrEF
Cardiac echography | 3 years
  Rest and low-effort evaluation of cardiac parameters
Cardiac calcium scoring | 3 years
  Evaluation of calcium scoring among participants
Cardiac MRI | 3 years
  Novel biomarkers of cardiac fibrosis, extra-cellular volume, matrix remodeling
Left atria | 3 years
  Evaluation of LA remodeling (volumes) and function (strain)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien HULOT, MD PhD, Principal Investigator — AP - HP, Hôpital Européen Georges-Pompidou, Paris, France
Locations (1):
- AP - HP, Hôpital Européen Georges-Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data used for publication could be shared through scientific collaboration with the sponsor or any collaborations implied.The sharing will respect the unital consortium agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Will become available from the time when summary data are published
Access Criteria: Sharing access criteria will be discussed between the sponsor and collaborate

REFERENCES:
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] De Peretti, et al. Prévalence et statut fonctionnel des cardiopathies ischémiques et de l'insuffisance cardiaque dans la population adulte en France : apports des enquêtes déclaratives " Handicap-Santé " BEH 2014; (9-10):172-81
- [Background] Galinier M, et al. Parcours de Soins. Dossier insuffisance cardiaque, encore trop d'hospitalisations pourtant évitables. État des lieux en France en 2013. Le Concours Médical 2013; 135(6):443-7
- [Background] Lindenfeld J, Albert NM, Boehmer JP et coll. HFSA 2010 Comprehensive Heart Failure Practice Guideline. J Card Fail 2010 ; 16 (6): e1-e194. - Arnold JM, Liu P, Demers C et coll. Canadian Cardiovascular Society consensus conference recommendations on heart failure 2006: diagnosis and management. Can J Cardiol 2006 ; 22 (1) : 23-45
- [Background] Blanc - SVSE 1 - Physiologie, physiopathologie, santé publique (Blanc SVSE 1) 2013
- [Background] Vasan RS, Levy D. The role of hypertension in the pathogenesis of heart failure. A clinical mechanistic overview. Arch Intern Med. 1996 Sep 9;156(16):1789-96. PMID 8790072
- [Background] Fonarow GC, Stough WG, Abraham WT, Albert NM, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Hospitals. Characteristics, treatments, and outcomes of patients with preserved systolic function hospitalized for heart failure: a report from the OPTIMIZE-HF Registry. J Am Coll Cardiol. 2007 Aug 21;50(8):768-77. doi: 10.1016/j.jacc.2007.04.064. Epub 2007 Aug 6. PMID 17707182
- [Background] CDC statistics 2016; AHA Heart disease and stoke statistics 2017; European CVD statistics 2017 ; Dunlay S et al 2017 Nat Rev Cardiol
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Zile MR, Gottdiener JS, Hetzel SJ, McMurray JJ, Komajda M, McKelvie R, Baicu CF, Massie BM, Carson PE; I-PRESERVE Investigators. Prevalence and significance of alterations in cardiac structure and function in patients with heart failure and a preserved ejection fraction. Circulation. 2011 Dec 6;124(23):2491-501. doi: 10.1161/CIRCULATIONAHA.110.011031. Epub 2011 Nov 7. PMID 22064591
- [Background] Katz DH, Beussink L, Sauer AJ, Freed BH, Burke MA, Shah SJ. Prevalence, clinical characteristics, and outcomes associated with eccentric versus concentric left ventricular hypertrophy in heart failure with preserved ejection fraction. Am J Cardiol. 2013 Oct 15;112(8):1158-64. doi: 10.1016/j.amjcard.2013.05.061. Epub 2013 Jun 28. PMID 23810323
- [Background] Lam CS, Roger VL, Rodeheffer RJ, Bursi F, Borlaug BA, Ommen SR, Kass DA, Redfield MM. Cardiac structure and ventricular-vascular function in persons with heart failure and preserved ejection fraction from Olmsted County, Minnesota. Circulation. 2007 Apr 17;115(15):1982-90. doi: 10.1161/CIRCULATIONAHA.106.659763. Epub 2007 Apr 2. PMID 17404159
- [Background] Persson H, Lonn E, Edner M, Baruch L, Lang CC, Morton JJ, Ostergren J, McKelvie RS; Investigators of the CHARM Echocardiographic Substudy-CHARMES. Diastolic dysfunction in heart failure with preserved systolic function: need for objective evidence:results from the CHARM Echocardiographic Substudy-CHARMES. J Am Coll Cardiol. 2007 Feb 13;49(6):687-94. doi: 10.1016/j.jacc.2006.08.062. Epub 2007 Jan 26. PMID 17291934
- [Background] Shah AM, Claggett B, Kitzman D, Biering-Sorensen T, Jensen JS, Cheng S, Matsushita K, Konety S, Folsom AR, Mosley TH, Wright JD, Heiss G, Solomon SD. Contemporary Assessment of Left Ventricular Diastolic Function in Older Adults: The Atherosclerosis Risk in Communities Study. Circulation. 2017 Jan 31;135(5):426-439. doi: 10.1161/CIRCULATIONAHA.116.024825. Epub 2016 Dec 7. PMID 27927714
- [Background] Borbely A, van der Velden J, Papp Z, Bronzwaer JG, Edes I, Stienen GJ, Paulus WJ. Cardiomyocyte stiffness in diastolic heart failure. Circulation. 2005 Feb 15;111(6):774-81. doi: 10.1161/01.CIR.0000155257.33485.6D. Epub 2005 Feb 7. PMID 15699264
- [Background] van Heerebeek L, Borbely A, Niessen HW, Bronzwaer JG, van der Velden J, Stienen GJ, Linke WA, Laarman GJ, Paulus WJ. Myocardial structure and function differ in systolic and diastolic heart failure. Circulation. 2006 Apr 25;113(16):1966-73. doi: 10.1161/CIRCULATIONAHA.105.587519. Epub 2006 Apr 17. PMID 16618817
- [Background] Zile MR, Baicu CF, Ikonomidis JS, Stroud RE, Nietert PJ, Bradshaw AD, Slater R, Palmer BM, Van Buren P, Meyer M, Redfield MM, Bull DA, Granzier HL, LeWinter MM. Myocardial stiffness in patients with heart failure and a preserved ejection fraction: contributions of collagen and titin. Circulation. 2015 Apr 7;131(14):1247-59. doi: 10.1161/CIRCULATIONAHA.114.013215. Epub 2015 Jan 30. PMID 25637629
- [Background] Adeniran I, MacIver DH, Hancox JC, Zhang H. Abnormal calcium homeostasis in heart failure with preserved ejection fraction is related to both reduced contractile function and incomplete relaxation: an electromechanically detailed biophysical modeling study. Front Physiol. 2015 Mar 20;6:78. doi: 10.3389/fphys.2015.00078. eCollection 2015. PMID 25852567
- [Background] van Heerebeek L, Hamdani N, Falcao-Pires I, Leite-Moreira AF, Begieneman MP, Bronzwaer JG, van der Velden J, Stienen GJ, Laarman GJ, Somsen A, Verheugt FW, Niessen HW, Paulus WJ. Low myocardial protein kinase G activity in heart failure with preserved ejection fraction. Circulation. 2012 Aug 14;126(7):830-9. doi: 10.1161/CIRCULATIONAHA.111.076075. Epub 2012 Jul 17. PMID 22806632
- [Background] Rommel KP, von Roeder M, Latuscynski K, Oberueck C, Blazek S, Fengler K, Besler C, Sandri M, Lucke C, Gutberlet M, Linke A, Schuler G, Lurz P. Extracellular Volume Fraction for Characterization of Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2016 Apr 19;67(15):1815-1825. doi: 10.1016/j.jacc.2016.02.018. PMID 27081022
- [Background] Mohammed SF, Hussain S, Mirzoyev SA, Edwards WD, Maleszewski JJ, Redfield MM. Coronary microvascular rarefaction and myocardial fibrosis in heart failure with preserved ejection fraction. Circulation. 2015 Feb 10;131(6):550-9. doi: 10.1161/CIRCULATIONAHA.114.009625. Epub 2014 Dec 31. PMID 25552356
- [Background] Kjekshus J, Apetrei E, Barrios V, et al. Rosuvastatin in older patients with systolic heart failure. N Engl J Med 2007;357:2248-61. / Weber T, Auer J, O'Rourke MF, et al. Prolonged mechanical systole and increased arterial wave reflections in diastolic dysfunction. Heart 2006;92:1616-22 / Desai AS, Mitchell GF, Fang JC, et al. Central aortic stiffness is increased in patients with heart failure and preserved ejection fraction. J Card Fail 2009;15:658-64.
- [Background] Lam CS, Roger VL, Rodeheffer RJ, Borlaug BA, Enders FT, Redfield MM. Pulmonary hypertension in heart failure with preserved ejection fraction: a community-based study. J Am Coll Cardiol. 2009 Mar 31;53(13):1119-26. doi: 10.1016/j.jacc.2008.11.051. PMID 19324256
- [Background] Kenchaiah S, Evans JC, Levy D, et al. Obesity and the risk of heart failure. N Engl J Med 2002; 347:305-13 / Ebong IA, Goff DC Jr., Rodriguez CJ, et al. The relationship between measures of obesity and incident heart failure: the multi-ethnic study of atherosclerosis. Obesity (Silver Spring) 2013;21: 1915-22 / Sundström J, Bruze G, Ottosson J, et al. Weight loss and heart failure: a nationwide study of gastric bypass surgery versus intensive lifestyle treatment. Circulation 2017;135:1577-85.
- [Background] Lainscak M, Anker SD. Heart failure, chronic obstructive pulmonary disease, and asthma: numbers, facts, and challenges. ESC Heart Fail. 2015 Sep;2(3):103-107. doi: 10.1002/ehf2.12055. Epub 2015 Jul 31. PMID 27708851
- [Background] Ather S, Chan W, Bozkurt B, Aguilar D, Ramasubbu K, Zachariah AA, Wehrens XH, Deswal A. Impact of noncardiac comorbidities on morbidity and mortality in a predominantly male population with heart failure and preserved versus reduced ejection fraction. J Am Coll Cardiol. 2012 Mar 13;59(11):998-1005. doi: 10.1016/j.jacc.2011.11.040. PMID 22402071
- [Background] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313
- [Background] Villemain O, Correia M, Mousseaux E, Baranger J, Zarka S, Podetti I, Soulat G, Damy T, Hagege A, Tanter M, Pernot M, Messas E. Myocardial Stiffness Evaluation Using Noninvasive Shear Wave Imaging in Healthy and Hypertrophic Cardiomyopathic Adults. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1135-1145. doi: 10.1016/j.jcmg.2018.02.002. Epub 2018 Mar 14. PMID 29550319
- [Derived] Raboudi A, Herve PY, Allanic M, Boutinaud P, Christophe JJ, Firat H, Mousseaux E, Pernot M, Prot P, Sartorius-Carvajal A, Chezalviel-Guilbert F, Hulot JS; PACIFIC consortium. The PACIFIC ontology for heterogeneous data management in cardiology. J Biomed Inform. 2024 Jan;149:104579. doi: 10.1016/j.jbi.2023.104579. Epub 2023 Dec 20. PMID 38135173
- [Derived] Raboudi A, Allanic M, Balvay D, Herve PY, Viel T, Yoganathan T, Certain A, Hilbey J, Charlet J, Durupt A, Boutinaud P, Eynard B, Tavitian B. The BMS-LM ontology for biomedical data reporting throughout the lifecycle of a research study: From data model to ontology. J Biomed Inform. 2022 Mar;127:104007. doi: 10.1016/j.jbi.2022.104007. Epub 2022 Feb 4. PMID 35124236